CLINICAL TRIAL: NCT05765734
Title: A Phase 1/2 Study of TAS3351 in Patients With Advanced Non-Small Cell Lung Cancer and EGFR Mutations
Brief Title: A Study of TAS3351 in NSCLC Patients With EGFRmt
Acronym: TAS3351
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic decision, not based on safety concerns
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10073010; 2022-502595-23 (EudraCT Number)
Record Dates: First submitted 2023-02-08; First posted 2023-03-13 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; EGFR mutation; C797S mutation; TAS3351
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAS3351 Part A (Dose Escalation) (Experimental): Dose escalation will assess the safety and determine the recommended phase 2 dose and regimen of TAS3351 administered orally.
  Interventions: Drug: TAS3351 oral administration
- TAS3351 Part B (Dose Expansion) (Experimental): TAS3351 in NSCLC patients with C797S EGFRmt. TAS3351 will be administered at the recommended phase 2 dose determined in Part A.
  Interventions: Drug: TAS3351 oral administration
- TAS3351 Part C (Phase 2) (Experimental): To assess efficacy of TAS3351 in NSCLC patients with C797S EGFRmt. TAS3351 will be administered at the recommended phase 2 dose.
  Interventions: Drug: TAS3351 oral administration

INTERVENTIONS:
Drug: TAS3351 oral administration — TAS3351 will be administered orally

SUMMARY:
This is a first-in-human, open label, Phase 1/2 study to investigate the safety and efficacy of TAS3351 in patients with advanced or metastatic non-small cell lung cancer (NSCLC) harboring an acquired C797S epidermal growth factor receptor (EGFR) mutation.

DETAILED DESCRIPTION:
This study will be conducted in 3 parts (i.e. dose escalation, dose expansion, and a phase 2 portion). The dose escalation part will investigate the safety and determine the recommended phase 2 dose and the recommended dosing regimen of TAS3351 administered orally. The dose expansion part will explore the efficacy of TAS3351 in NSCLC patients with C797S EGFR mutations. The phase 2 part will assess the efficacy of TAS3351 in NSCLC patients with C797S EGFR mutations.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, non-resectable or metastatic NSCLC
* Have adequate organ function
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Has tumor tissue available to allow for analysis of EGFRmt status

Dose Escalation:

• Has any EGFRmt status

Dose Escalation back-fill part, Dose Expansion and Phase II:

* Has any sensitizing EGFRmt and a confirmed C797S EGFRmt
* Has measurable disease per RECIST v1.1

Exclusion Criteria:

* Participating in medical research not compatible with this study
* Symptomatic and unstable CNS metastases
* Have not recovered from prior cancer treatment
* Have a significant cardiac condition
* Are a pregnant or breastfeeding female
* A serious illness or medical condition
* Unable to swallow or digest pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Dose Escalation: To investigate the safety and determine the recommended Phase 2 dose and dosing schedule of TAS3351 | baseline through cycle 1(each cycle is 21 days)
  Adverse Events
Dose Escalation: To investigate the safety and determine the recommended Phase 2 dose and dosing schedule of TAS3351 | baseline through cycle 1(each cycle is 21 days)
  Incidence of dose limiting toxicities (DLTs)
Dose Expansion: To explore the efficacy of TAS3351 | estimated 9 months
  Objective Response Rate (ORR)
Phase 2: To assess the efficacy of TAS3351 | estimated 3 years
  Objective Response Rate (ORR)

SECONDARY OUTCOMES:
Dose Escalation:To evaluate the antitumor activity of TAS3351 | estimated 20 months
  Objective response rate (ORR)
Dose Escalation:To evaluate the antitumor activity of TAS3351 | estimated 20 months
  Duration of response (DoR)
Dose Escalation:To evaluate the antitumor activity of TAS3351 | estimated 20 months
  Disease control rate (DCR)
Dose Escalation: To evaluate the antitumor activity of TAS3351 | estimated 20 months
  Progression free survival (PFS)
Dose Escalation: To evaluate the antitumor activity of TAS3351 | estimated 20 months
  Overall Survival (OS)
Dose Escalation: To characterize the pharmacokinetics (PK) of TAS3351 | Cycle 1 Day 1 through cycle 1 Day 15 (21-Day cycle)
  Evaluate the maximum plasma concentration (Cmax)
Dose Escalation: To characterize the pharmacokinetics (PK) of TAS3351 | ECycle 1 Day 1 through cycle 1 Day 15 (21-Day cycle)
  Area under the plasma concentration-time curve (AUC)
Dose Expansion: To confirm the safety and tolerability of TAS3351 at the recommended phase 2 dose and dosing schedule | estimated 9 months
  Adverse Events (AEs)
Dose Expansion: To further explore the anti-tumor efficacy of TAS3351 | estimated 9 months
  Duration of response (DoR) by ICR
Dose Expansion: To further explore the anti-tumor efficacy of TAS3351 | estimated 9 months
  Progression Free Survival (PFS) by ICR
Dose Expansion: To further explore the anti-tumor efficacy of TAS3351 | estimated 9 months
  Disease Control Rate (DCR) by ICR
Dose Expansion: To further explore the anti-tumor efficacy of TAS3351 | estimated 9 months
  Objective Response Rate (ORR) by Investigator Assessment
Dose Expansion: To further explore the anti-tumor efficacy of TAS3351 | estimated 9 months
  Duration of Response (DoR) by Investigator Assessment
Dose Expansion: To further explore the anti-tumor efficacy of TAS3351 | estimated 9 months
  Progression Free Survival (PFS) by Investigator Assessment
Dose Expansion: To further explore the anti-tumor efficacy of TAS3351 | estimated 9 months
  Disease Control Rate (DCR) by Investigator Assessment
Dose Expansion: To further explore the anti-tumor efficacy of TAS3351 | estimated 9 months
  Intracranial Objective Response Rate (icORR)
Dose Expansion: To further explore the anti-tumor efficacy of TAS3351 | estimated 9 months
  Intracranial Duration of Response (icDOR)
Dose Expansion: To further explore the anti-tumor efficacy of TAS3351 | estimated 9 months
  Overall survival (OS)
Phase 2: To evaluate the safety and tolerability of TAS3351 | estimated 3 years
  Adverse Events (AEs)
Phase 2: To further assess the efficacy of TAS3351 | estimated 3 years
  Duration of response (DoR) by ICR
Phase 2: To further assess the efficacy of TAS3351 | estimated 3 years
  Progression Free Survival (PFS) by ICR
Phase 2: To further assess the efficacy of TAS3351 | estimated 3 years
  Disease Control Rate (DCR) by ICR
Phase 2: To further assess the efficacy of TAS3351 | estimated 3 years
  Objective Response Rate (ORR) by Investigator Assessment
Phase 2: To further assess the efficacy of TAS3351 | estimated 3 years
  Duration of Response (DoR) by Investigator Assessment
Phase 2: To further assess the efficacy of TAS3351 | estimated 3 years
  Progression Free Survival (PFS) by Investigator Assessment
Phase 2: To further assess the efficacy of TAS3351 | estimated 3 years
  Disease Control Rate (DCR) by Investigator Assessment
Phase 2: To further assess the efficacy of TAS3351 | estimated 3 years
  Intracranial Objective Response Rate (icORR)
Phase 2: To further assess the efficacy of TAS3351 | estimated 3 years
  Intracranial Duration of Response (icDOR)
Phase 2: To further assess the efficacy of TAS3351 | estimated 3 years
  Overall survival (OS)
Phase 2:To evaluate patient reported outcomes (PROs) | estimated 3 years
  responses to patient questionnaires

CONTACTS AND LOCATIONS:
Locations (17):
- United States (4):
  - Georgetown University - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - Next Oncology - Virginia, Fairfax, Virginia
- Institut Gustave Roussy, Villejuif, Val De Marne, France
- Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia, Germany
- IEO Istituto Europeo di Oncologia, Milan, Italy
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - Cancer Institute Hospital of JFCR, Kōtoku
- Netherlands (2):
  - Antoni van Leeuwenhoek, Amsterdam
  - Leiden University Medical Center (LUMC), Leiden
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- The Christie Hospital, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No